CLINICAL TRIAL: NCT04952246
Title: Clinical Isolated Spinal Cord Syndrome Was Identified as Multiple Sclerosis Associated Risk Factor Analysis
Brief Title: Clinical Isolation Syndrome of Spinal Cord and Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020513
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Clinical Isolation Syndrome of Spinal Cord; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis group
- non-prognosis group

SUMMARY:
The purpose of this study was to investigate the factors that influence the progression of patients with clinically isolated spinal cord syndrome to multiple sclerosis.

DETAILED DESCRIPTION:
This study included patients who were first diagnosed with clinically isolated spinal cord syndrome admitted to the Department of Neurology, Peking University Third Hospital between January 2010 and November 2020. According to the result of the outcome is divided into multiple sclerosis and outcome group, analyzing the characteristics of the age, sex, clinical manifestations, imaging features, evoked potential, blood immune antibody results, rate of cerebrospinal fluid routine biochemical synthesis oligoclonal band IgG, extension, nerve dysfunction score spinal cord clinically isolated syndrome and the influence factors, such as the relationship between the outcome of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis time and place: Department of Neurology, Peking University Third Hospital from January 2010 to November 2020 Diagnosed as a patient with clinically isolated spinal cord syndrome for the first time

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: clinically isolated spinal cord syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Progressed to multiple sclerosis | 3 years
  Progressed to multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijin, China